CLINICAL TRIAL: NCT03214848
Title: Evaluation of an Intervention to Increase Post-abortion LARC Uptake: A Randomized Controlled Trial of Educational and Financial Counseling Prior to Clinical Presentation.
Brief Title: Evaluation of an Intervention to Increase Post-abortion LARC Uptake.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Woodruff Health Sciences Center Foundation (Unknown)
Responsible Party: Principal Investigator, Lisa Haddad, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB00094882
Record Dates: First submitted 2017-07-10; First posted 2017-07-12 (Actual); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Post Abortion Contraception
Keywords: Long-acting reversible contraceptive; Post Abortion; Iintrauterine device; Contraceptive implant; LARC; IUD

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standart of Care (No Intervention): Standard of care at the clinic is to discuss the abortion procedure without specific contraceptive counseling given prior to the day of abortion procedure.
- Contraceptive education prior to abortion (Experimental): Addition (to the standard or care) of a brief phone contraceptive education with optional financial counseling referral prior to abortion visit.
  Interventions: Behavioral: Contraceptive education prior to abortion

INTERVENTIONS:
Behavioral: Contraceptive education prior to abortion — Contraceptive education script will be delivered over the phone prior to abortion visit.
  Arms: Contraceptive education prior to abortion

SUMMARY:
This is a randomized prospective study evaluating the impact of a brief contraceptive education intervention with optional referral for financial counseling on post abortion long-acting reversible contraceptive (LARC) uptake and contraceptive use at three months post abortion.

DETAILED DESCRIPTION:
As repeat unintended pregnancy and abortion remain public health challenges, increasing long-acting reversible contraceptive (LARC), specifically intrauterine device (IUD) and contraceptive implant, use among women presenting for abortion care is a priority. Despite its efficacy and safety, LARC methods remain underutilized in the abortion setting.

This is a randomized prospective study evaluating the impact of a brief contraceptive education intervention with optional referral for financial counseling on post abortion long-acting reversible contraceptive (LARC) uptake and contraceptive use at three months post abortion.

ELIGIBILITY:
Inclusion Criteria:

* Women calling to schedule an appointment for an abortion and/or those who receive abortion services at the Atlanta Women's Center with fluency in English and able to provide informed consent
* 16 years and older

Exclusion Criteria:

-Younger than 16 years old

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 1314 (Actual)
Dates: Start 2017-09-13 (Actual); Primary Completion 2018-02-21 (Actual); Study Completion 2018-02-21 (Actual)

PRIMARY OUTCOMES:
Proportion of Long-Acting Reversible Contraception (LARC) methods inserted immediately post abortion in the intervention and standard of care arms. | Immidiately post abortion (day of the procedure).
  Proportion of LARC methods inserted immediately post abortion in the intervention and standard of care arms will be calculated based on data abstracted from patients' medical records.

SECONDARY OUTCOMES:
Proportion of Long-Acting Reversible Contraception (LARC) methods used in the intervention and standard of care arms three months post abortion. | Three months post abortion.
  This outcome is inclusive of immediate initiators and those who initiate by three months. Proportion of LARC methods used in the intervention and standard of care arms will be calculated based on the 3-month follow-up phone interview.
Cost-effectiveness analysis of the study intervention. | Three months post abortion.
  The cost-effectiveness analysis will involve multiple parts. The study team will initially complete a cost description of the interventions involving time spent in developing the scripts for LARC education and financial counseling, and additional time spent making contact with women and providing the augmented counseling compared to the initial pre-communication session.Incremental cost-effectiveness ratios for the intervention overall will be calculated compared to a 'base-case' of standard of care in the primary analysis. This value will provide cost per additional women using LARC. In a secondary analysis, the study team will compare differences between women receiving the educational component only versus 'base-case', and also women receiving the educational and financial counseling component versus 'base-case'.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Haddad, MD, Principal Investigator — Emory University
Locations (1):
- Atlanta Women's Center, Atlanta, Georgia, United States